CLINICAL TRIAL: NCT06273553
Title: An Open-Label, Phase 1/2 Study to Evaluate the Safety, Tolerability, Immunogenicity and Efficacy of RG002 Injection (an mRNA Therapeutic Vaccine) in Subjects With Human Papillomavirus (HPV) 16 or 18 Associated Cervical Intraepithelial Neoplasia Grade 2 or 3 (CIN2/3)
Brief Title: A Study in Subjects With Human Papillomavirus 16 or 18 Associated Cervical Intraepithelial Neoplasia Grade 2 or 3
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RinuaGene Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG002-A1201
Record Dates: First submitted 2024-01-31; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Human Papillomavirus Associated Intraepithelial Neoplasia; Cervical Intraepithelial Neoplasia Grade 2/3; Human Papillomavirus Type 16 Infection; Human Papillomavirus Type 18 Infection
Keywords: HPV 16 or 18; mRNA vaccine; CIN 2; CIN 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RG002 Injection (Experimental): In Part A, subjects with histologically confirmed Cervical Intraepithelial Neoplasia Grade 2 or 3 (CIN2/3) associated with Human Papillomavirus (HPV) 16 or 18, will be allocated to three dose cohorts that are 25µg,75µg and 150µg. In Part B, subjects with histologically confirmed Cervical Intraepithelial Neoplasia Grade 2 or 3 (CIN2/3) associated with Human Papillomavirus (HPV) 16 or 18, will be allocated to 1 or 2 dose levels according to the results of Part A. All subjects will receive a total of three RG002 Injections, administered intramuscularly at assigned dose level, with a dosing frequency of every 2 weeks (D1, D15, and D29).
  Interventions: Biological: RG002 injection

INTERVENTIONS:
Biological: RG002 injection — In Part A, there are three dose cohorts that are 25µg,75µg and 150µg. In Part B, there will 1 or 2 dose levels according to the results of Part A. All subjects will receive a total of three RG002 Injections, administered intramuscularly at assigned dose level, with a dosing frequency of every 2 weeks (D1, D15, and D29).

SUMMARY:
The purpose of this study is to to evaluate the safety, tolerability, immunogenicity, and efficacy of RG002 Injection in subjects with HPV16/18 associated Cervical Intraepithelial Neoplasia Grade 2 or 3(CIN2/3).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with study site guidelines.
2. Female 18~45 years of age when signing the ICF for Part A, and 18~55 years of age when signing the ICF for Part B.
3. Body mass index (BMI) ≤30 kg/m2.
4. Pathological diagnosis of CIN Grade 2 or 3 as confirmed by central pathological reviewers within 12 weeks prior to administration of first study vaccination.
5. The lesion of CIN Grade 2 or 3 is large enough for histopathologic biopsy at screening and during treatment.
6. Has a satisfactory colposcopy at screening, i.e., the entire lesion as well as the entire squamocolumnar junction (type 1 or 2 transformation zone) is visualizable by colposcopy;
7. Confirmed high-risk HPV infection with HPV16+ and / or HPV18+ by a commercially available high-risk DNA assay (e.g., Cobas® HPV test from Roche).
8. Adequate hematologic, renal, and hepatic function are determined by the Investigator, based upon medical history, physical examination, and laboratory test results at screening:

   1. Bone marrow function: absolute neutrophil count ≥1,500/µL, hemoglobin (HGB) ≥ 9 g/dL, and platelets ≥ 100,000/ µL.
   2. Renal function: creatinine ≤ 1.5 × institutional upper limit of normal (ULN).
   3. Hepatic function: total bilirubin ≤ 1.5 × ULN, Aspartate aminotransferase (AST) and/or alanine transaminase (ALT) ≤ 1.5 × ULN.
9. Women of child-bearing potential (WOCBP) agree to remain sexually abstinent, use medically effective contraception (i.e., complex contraception, male condom and spermicide, contraceptive patches, barrier methods, spermicide, etc.), from enrollment to 9 months after the last injection or have a partner who is sterile (i.e., vasectomy).
10. Able and willing to comply with all study procedures.

Exclusion Criteria:

1. Cervical adenocarcinoma in situ (AIS), or atypical endometrial or glandular cells, or evidence of invasive cervical carcinoma on cervical biopsy within 12 weeks prior to administration of first study vaccination.
2. High-grade intraepithelial neoplasia or invasive carcinoma of vulva, vagina or anus.
3. History of severe allergy to any vaccine or serious hypersensitivity reaction to a known ingredient (e.g., PEG) of RG002 injection judged by the investigator.
4. Active infection with herpes simplex virus (HSV).
5. Positive serological test at screening for HIV virus, active syphilis infection, or positive hepatitis B virus surface antigen (HbsAg) and the number of copies of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) ≥ 500 IU/mL (or 2500 copies, or the lower limit of the positive detection value of the study site) at screening, or HbsAg (-), hepatitis B core antibody (HbcAb) (+) and the number of copies of HBV DNA ≥ 500 IU/mL (or 2500 copies, or the lower limit of the positive detection value of the study site) after treatment of HBV infection, or positive hepatitis C antibody (HCV-Ab) and hepatitis C virus (HCV) ribonucleic acid (RNA) ≥ ULN of the study site.
6. Subjects with a concurrent condition of fatty liver disease at screening.
7. Subjects with poorly controlled diabetes (fasting blood glucose ≥ 10mmol/L) after drug treatment at screening.
8. History of serious cardiovascular and cerebrovascular diseases, including but not limited to serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention; repeated 12-lead ECG with QTcF interval ≥ 470 msec; acute coronary syndrome, congestive cardiac failure, aortic dissection, stroke or other Grade 3 or above cardiovascular and cerebrovascular events within 6 months before the first administration; New York Heart Association (NYHA) cardiac function classification ≥ Grade III or hypertension that cannot be clinically controlled (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg).
9. Major surgery (except for surgery for diagnostic purposes) within 4 weeks before the first administration or expected to undergo major surgery (except for surgery for diagnostic purposes) during the study period; If major surgery occurred > 4 weeks prior to the first administration of the study, individual must have recovered adequately from the toxicity and/or complications from the intervention prior to the first administration of the study.
10. Hereditary hemorrhagic tendency or coagulation dysfunction, or a history of thrombosis or hemorrhagic disease, or requirement of continuous use of anticoagulants.
11. Female subjects in pregnancy or lactation, or a positive result on a serum human chorionic gonadotropin (HCG) test at screening (Visit 1) or a positive urine pregnancy test pre-vaccination at Visit 2 (and at subsequent vaccination visits).
12. Currently receiving or has received treatment with systemic steroids in the following dosages prior to administration of the first study vaccination.

    1. Long-term corticosteroids: ≥0.5 mg/kg/day of oral prednisolone or equivalent, within 30 days prior to administration of the first study vaccination.
    2. Sporadic corticosteroids: ≥1 mg/kg/day of oral prednisolone or equivalent for 2 or more short courses of > 3 days.

    Note: Current or recent use of eye drop or inhaled glucocorticoid therapy is acceptable.
13. Immunosuppression due to treatment for concurrent disease or medical history: HIV treatment, antirheumatic drugs, organ or bone marrow transplantation or relevant treatment.
14. Systemic treatment for malignancy within 2 years of enrollment.
15. Administration of any blood product within 3 months of enrollment.
16. Administration of any vaccine within 4 weeks of enrollment.
17. A history of any therapeutic HPV vaccination (commercially approved prophylactic HPV vaccination is acceptable).
18. Other condition or prior therapy that, in the opinion of the investigator, compromises the subject's welfare or may confound study results.
19. Tattoos, scars, or active lesions/rashes within 2 cm of the intended site of vaccination (deltoid muscle) or any implantable leads, that may affect the safety observation.
20. Adverse events that do not recover to grade 1 during the screening period.
21. Subjects are currently participating or has participated in a study with an investigational drug or device within 30 days of signing informed consent.
22. Subjects who are judged by the investigator to have a history of other serious systemic diseases, or not suitable for participating in the trial for any other reason (the subject has mental illness, alcohol abuse, drug use or drug abuse that may affect her compliance with the trial or may interfere with the interpretation of the study results).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability of RG002 Injection, measured by the incidence of adverse events | Week 9
  Safety and Tolerability of RG002 Injection will be measured by the incidence of adverse events per CTCAE v5.0
Part A: Maximum tolerated dose (MTD) and/or RP2D of RG002 Injection | MTD:Week 9; RP2D: Week 36
Part B: Primary efficacy of RG002 Injection, measured by the proportion of subjects with histopathological regression | Week36
  The proportion of subjects with histopathological regression to either CIN1 or normal at Week 36

SECONDARY OUTCOMES:
Part A: Preliminary efficacy of RG002 Injection,measured by proportion of subjects with histopathological regression | Week36
  The proportion of subjects with histopathological regression to either CIN1 or normal at Week 36
Part A: Preliminary efficacy of RG002 Injection,measured by proportion of subjects with clearance of HPV16/18 | Week36
  The clearance of HPV16 or HPV18 will be evaluated according to the results of HPV test at Week 21 and Week 36.
Part A: Preliminary efficacy of RG002 Injection,measured by proportion of subjects with histopathological regression and clearance of HPV16/18 | Week36
  The proportion of subjects with histopathological regression to CIN1 or normal and clearance of HPV16 or HPV18, or both at Week36.
Part A and B: Immunogenicity of RG002 Injection,measured by the level of cellular immune response | Week36
  The level of cellular immune response in Peripheral blood mononuclear cells (PBMCs) as measured by IFN-γ enzyme-linked immunosorbent spot-forming (ELISpot) assay
Part A and B: Immunogenicity of RG002 Injection,measured by the proportion of T lymphocytes | Week36
  The immuno-phenotyping including the proportion of CD3+CD4+CD137+ and CD3+CD8+CD137+ T lymphocytes in whole blood as measured by flow cytometry.
Part A and B: Immunogenicity of RG002 Injection,measured by the expression of cytokines in serum | Week36
  The expression of cytokines in serum, i.e., IL-1β, IL-1ra, IL-2, IL-6, IL-10, GM-CSF, TNF-α and IFN-γ measured by MSD® Assays.
Part A and B: Immunogenicity of RG002 Injection,measured by the serum levels of anti-HPV16 and anti-HPV18 IgG antibodies. | Week36
  Serum levels of anti-HPV16 and anti-HPV18 IgG antibodies as measured by Luminex.
Part A and B: Exposure level of RG002 Injection, measured by mRNA | Week7
  The plasma exposure level(AUC, Cmax, etc.) of mRNA will be measured Real Time Quantitative-Polymerase Chain Reaction (RT-qPCR)
Part A and B: Exposure level of RG002 Injection, measured by cationic lipids | Week7
  The plasma exposure level(AUC, Cmax, etc.) of cationic lipids will be measured by Liquid Chromatography Tandem Mass Spectrometry(LC-MS/MS).
Part A and B: Anti-drug antibody (ADA) to polyethylene glycol (PEG) of RG002 injection, measured by the serum titer of anti-PEG IgG and anti-PEG IgM | Week6
  The serum titer of anti-PEG IgG and anti-PEG IgM as measured by enzyme-linked immunosorbent assay (ELISA).
Part B: Secondary efficacy, measured by proportion of subjects with histopathological regression | Week36
  The proportion of subjects with histopathological regression to either CIN1 or normal at Week 36
Part B: Secondary efficacy, measured by proportion of subjects with clearance of HPV16/18 | Week36
  The clearance of HPV16 or HPV18 will be evaluated according to the results of HPV test at Week 21 and Week 36.
Part B: Secondary efficacy, measured by proportion of subjects with histopathological regression and clearance of HPV16/18 | Week36
  The proportion of subjects with histopathological regression to CIN1 or normal and clearance of HPV16 or HPV18, or both at Week36.
Part B: Safety and tolerability of RG002 Injection, measured by the incidence of adverse events | Week9
  Safety and Tolerability of RG002 Injection will be measured by the incidence of adverse events per CTCAE v5.0
Part B: Optionally assess the biomarker of RG002 Injection, measured by the level of potential biomarkers and the level of infiltrating T cells and myeloid cells in the lesions. | Week36
  The level of potential biomarkers of RG002 Injection, i.e., CD45, CD3, CD4, CD8, CD25, FOXP3, PD-1, and CD137, and the level of infiltrating T cells (CD3, CD8, FOXP3, TIM3, Tbet, PD-1, DAPI) and myeloid cells (CD14, CD33, CD68, CD163, CD11c, PD-L1, DAPI) in the lesions.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338